CLINICAL TRIAL: NCT04802785
Title: The Impact of Air Travel on Passenger Cognitive Functions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dinara Zhumanbayeva (Other)
Responsible Party: Sponsor-Investigator, Dinara Zhumanbayeva, head of laboratory, lurye Clinic
Organization: lurye Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2021-02-17; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Air Travel
Keywords: Air Travel; health
MeSH Terms: interventions — Cytidine Diphosphate Choline; Cytochromes c6; Cytochromes c; Potassium Chloride; Sodium Citrate; Glucose; Domperidone; Simethicone; Aspirin; Magnesium Hydroxide; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The study Group (Experimental): 1. Before the flight in the conditions of the clinic's medical treatment room: Citicoline 500 mg(Vitaae®) and Cytochrome10 mg (Cytochrome C®) per os.
  2. 30 minutes before the flight: dilute 1 sachet of ORS® (Sodium Chloride 2.6 g+Potassium Chloride 1.5 g+Sodium Citrate 2.90 g+Dextrose 13.5 g) in 1 liter of water. Drink half of the solution (0.5 l) 30 minutes before the flight (at the airport). Also, 0.5 L of the solution will be provided on the plane during landing. If the flight lasts more than 1.5 hours, then dilute the second sachet of ORS® with 0.5-1 liters of water.
  3. 30 minutes before the flight (per os): Domperidone (Motilium ®) (1 tablet), Simethicone (Gas-X®) (3-4 capsules), Acetylsalicylic acid 150 mg and magnesium hydroxide 30,39 mg (Cardiomagnyl®)(1 tablet), probiotic (Bactistatin®) (1 capsule) per os.
  Interventions: Drug: Citicoline; Drug: Cytochrome C6; Drug: Sodium Chloride Oral Product; Drug: Potassium Chloride Oral Product; Drug: Sodium Citrate Oral Product; Drug: Dextrose Oral Tablet, Chewable; Drug: Domperidone Oral Product; Drug: Simethicone; Drug: Acetylsalicylic acid; Drug: Magnesium hydroxide; Drug: Probiotic Formula
- Control group (Active Comparator): Melatonin® 5 mg per os 2 hours before bedtime on the day of arrival for 3-4 days.
  Interventions: Drug: Melatonin 5 mg
- Explanatory group: (No Intervention): 12 participants without any intervention.

INTERVENTIONS:
Drug: Citicoline — Citicoline 500 mg (Vitaae®) per os
  Other Names: Citicoline (Vitaae®)
  Arms: The study Group
Drug: Cytochrome C6 — Cytochrome10 mg per os
  Other Names: (Cytochrome C®)
  Arms: The study Group
Drug: Sodium Chloride Oral Product — Sodium Chloride (NaCl) 2.6 g. per os
  Arms: The study Group
Drug: Potassium Chloride Oral Product — Potassium Chloride 1.5 g per os
  Other Names: Potassium Chloride
  Arms: The study Group
Drug: Sodium Citrate Oral Product — Sodium Citrate 2.90 g per os
  Other Names: Sodium Citrate
  Arms: The study Group
Drug: Dextrose Oral Tablet, Chewable — Dextrose 13.5 g per os
  Other Names: Dextrose
  Arms: The study Group
Drug: Domperidone Oral Product — Domperidone 1 tablet per os
  Other Names: Motilium ®
  Arms: The study Group
Drug: Simethicone — 3-4 capsules per os
  Other Names: Gas-X®
  Arms: The study Group
Drug: Acetylsalicylic acid — Acetylsalicylic acid 150 mg per os
  Arms: The study Group
Drug: Magnesium hydroxide — magnesium hydroxide 30 mg per os
  Arms: The study Group
Drug: Probiotic Formula — 1 capsule per os.
  Other Names: Bactistatin®
  Arms: The study Group
Drug: Melatonin 5 mg — Melatonin 5 mg per os.
  Other Names: Natrol Melatonin
  Arms: Control group

SUMMARY:
In the period from June 2021 to June 2022, a prospective clinical study will be conducted in the Republic of Kazakhstan with economy class passengers traveling by plane with a minimum flight period of 5-7 flight hours in the territory of the Republic of Kazakhstan.

ELIGIBILITY:
Study participants (Volunteers) will be recruited through media, advertisements and announcements. Prior to the study, study participants will receive written and oral explanations of the study protocols, and written informed consent will be obtained from each study participant. All potential research participants will undergo medical and psychological selection. The components, stages of selection are almost the same as those of general professional selection: the first stage is professiography / psychogram, the second stage is psychodiagnostics, the third stage is assessment and forecasting, and the fourth stage is decision making. Selection will assess the ability of participants to perform complex sequential actions.

Inclusion criterion:

* Age from 22 to 30 years old;
* at least 15 years of education, including secondary education;
* understand and speak Russian (Due to the valid Russian-language questionnaire and methodology).

In addition, study participants will be asked not to limit their caffeine intake from their daily intake, but only water is allowed 4 hours before the neuropsychological testing. Participants in the study should not hmedical/medicallane in the last two weeks prior to the start of the study, nor should they consume alcohol during the study.

Exclusion criterion:

* A member taking melatonin (affects circadian rhythm);
* Participant with comorbidities that affect cognitive function and sleep (eg, stroke, TIA, concussion with loss of consciousness, hearing problems, chronic fatigue syndrome, depression, seasonal affective disorder, anorexia);
* A participant with another ongoing sleep disorder.

All participants must be free of a history of venous thrombosis, antithrombotic or anticoagulant medications and oral contraceptives and / or any other drugs that interfere with blood coagulation (i.e. warfarin, coumadin) for at least 2 months prior to study initiation, and sign a consent to refrain from taking medications that may affect coagulation, such as aspirin or non-steroidal anti-inflammatory drugs, within 3 days after the flight, unless there is a medical / medical need.

-

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Urine Specific Gravity | 24 hours before the flight
  Urine Specific Gravity test
SpO2 level | 24 hours before the flight
  Pulse oximetry
Ultrasound examination | 24 hours before the flight
  Ultrasound examination of the veins of the lower limbs
The Liverpool Jet Lag questionnaire | 24 hours before the flight
  Changes from normal (0 to 5) while jetlag rating was recorded on a scale from 0 = insignificant jetlag to 10 = severe jetlag
Lake Louise Acute Mountain Sickness Assessment System | 24 hours before the flight
  Mild acute mountain sicknessas 3-5 points, moderate acute mountain sickness as 6-9 points, and severe acute mountain sickness as 10-12 points
Neuropsychological tests (Trail Making Test, Wechsler Memory Scale - IV, Free recall | 24 hours after the flight
  Word, color, and color-word T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal." In order for one score to be considered "higher" or "lower" than another, a 10 point or greater T score difference is required.

SECONDARY OUTCOMES:
The Liverpool Jet Lag questionnaire (LJLQ) | 24 hours after the flight
  Changes from normal (0 to 5) while jetlag rating was recorded on a scale from 0 = insignificant jetlag to 10 = severe jetlag
Lake Louise Acute Mountain Sickness Assessment System | 24 hours after the flight
  Mild acute mountain sicknessas 3-5 points, moderate acute mountain sickness as 6-9 points, and severe acute mountain sickness as 10-12 points
The Stroop Test | 24 hours after the flight
  Word, color, and color-word T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal." In order for one score to be considered "higher" or "lower" than another, a 10 point or greater T score difference is required.
Urine Specific Gravity | 24 hours after the flight
  Urine Specific Gravity test
SpO2 level | 24 hours before the flight
  Pulse oximetry

IPD SHARING:
Plan to Share IPD: No